CLINICAL TRIAL: NCT04133142
Title: Does Repetitive Peripheral Nerve Blocks Vs Single Peripheral Nerve Block Vs Standard Medical Treatment Provide a Better Pain Relief on Zoster Pain at the Acute Phase and Reduce the Risk of Post Herpetic Neuralgia?
Brief Title: Regional Anesthesia to Relief Zoster Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollement and covid
Sponsor: Vinmec Healthcare System (Other)
Responsible Party: Principal Investigator, Philippe Macaire, Anesthesiologist and Pain physician, Vinmec Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zona Blocks
Record Dates: First submitted 2019-10-11; First posted 2019-10-21 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Zoster Without Complications
Keywords: Zoster,; Pain relief; regional anesthesia; Prevention post herpetic neuralgia
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Intervention Model Description: Patient randomized in Medical treatment group or Early block group
  * medical treatment group will have standard pain medications and evaluation of pain relief at day 7
    * If pain reduce less or egal to VAS 4 medical treatment will continue it will be the control group
    * If no pain relief VAS more than 4 patient will be randomized to have
      * single block = Group late block single
      * or repeated blocks = Group late block repeated
  * ealy block group will be randomized to have
    * single block = Group early block single
    * or repeated blocks = Group early block repeated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Medical treatment (No Intervention): Patients receive the standard medical medication for herpes pain
  * Oral administration of Gabapentin
    * 300 mg/d on day 1 and 2
    * 600 mg/d on day 3 and 4 if pain persists
    * 900 mg/d on day 5 and 6 if pain persists
  * Oral administration of Paracetamol up to 3 g per day prescription for 7 day and continue for 3 weeks after evaluation
- Early block Single (Experimental): the patient will receive a regional anaesthesia by Inter fascial block, peripheral nerve block. Local anesthetic used will be ropivacaine 0.5% dose according to the type of block and never exceeding 3mg/kg The type of block would be the most appropriate to cover the dermatomes involved in the Herpes according to the mapping done with the higher ration benefit risks. Choice of Block by an anesthesiologist expert in regional anaesthesia techniques. After the block performance if the pain comes back patient will receive the standard medical treatment as in the group medical treatment
  Interventions: Procedure: peripheral nerve block, inter fascial nerve block
- Early Repeated block (Experimental): the patient will receive a regional anaesthesia by Inter fascial block, peripheral nerve block. The type of block would be the most appropriate to cover the dermatomes involved in the Herpes according to the mapping done with the higher ratio benefit risks. Local anesthetic used will be ropivacaine 0.5% dose according to the type of block and never exceeding 3mg/kg The choice of the block will be done by an anesthesiologist expert in regional anaesthesia techniques. The block will be repeated every 48h until the pain will reach VAS < 3 6 h after block recovery.
  Interventions: Procedure: peripheral nerve block, inter fascial nerve block
- Late block single (Experimental): Patients receive the standard medical medication for herpes pain
  * Oral administration of Gabapentin
    * 300 mg/d on day 1 and 2
    * 600 mg/d on day 3 and 4 if pain persists
    * 900 mg/d on day 5 and 6 if pain persists
  * Oral administration of Paracetamol up to 3 g per day at day 7 if pain more than VAS 4 the patient will receive a regional anaesthesia by Inter fascial block, peripheral nerve block . Local anesthetic used will be ropivacaine 0.5% dose according to the type of block and never exceeding 3mg/kg The type of block would be the most appropriate to cover the dermatomes involved in the Herpes according to the mapping done with the higher ration benefit risks. Choice of Block by an anesthesiologist expert in regional anaesthesia techniques. After the block performance if the pain comes back patient will receive the standard medical treatment as in the group medical treatment
  Interventions: Procedure: peripheral nerve block, inter fascial nerve block
- late block repeated (Experimental): Patients receive the standard medical medication for herpes pain
  * Oral administration of Gabapentin
    * 300 mg/d on day 1 and 2
    * 600 mg/d on day 3 and 4 if pain persists
    * 900 mg/d on day 5 and 6 if pain persists
  * Oral administration of Paracetamol up to 3 g per day prescription for 7 day and continue for 3 weeks after evaluation At day 7 if pain more than VAS 4 the patient will receive a regional anaesthesia by Inter fascial block, peripheral nerve block. The type of block would be the most appropriate to cover the dermatomes involved in the Herpes according to the mapping done with the higher ratio benefit risks. Local anesthetic used will be ropivacaine 0.5% dose according to the type of block and never exceeding 3mg/kg The choice of the block will be done by an anesthesiologist expert in regional anaesthesia techniques. The block will be repeated every 48h until the pain will reach VAS < 3 6 h after block recovery.
  Interventions: Procedure: peripheral nerve block, inter fascial nerve block

INTERVENTIONS:
Procedure: peripheral nerve block, inter fascial nerve block — regional anaesthesia by Inter fascial block, peripheral nerve block. The type of block would be the most appropriate to cover the dermatomes involved in the Herpes according to the mapping done with the higher ratio benefit risks. The choice of the block will be done by an anesthesiologist expert in regional anaesthesia techniques. local anesthetic will be ropivacaine 0.5% posology according to the type of block
  Arms: Early Repeated block; Early block Single; Late block single; late block repeated

SUMMARY:
Pain in Herpes is a serious issue for patients. at the acute phase it is a moderate to severe pain . 30% patients will develop a post herpetic neuralgia this percentage up to 70 % after 60 years old. this post herpetic neuralgia will affect their life. Publication showed the efficiency of regional anesthesia on pain at the acute phase and a recent meta-analysis showed the role of efficient pain relief on the prevention of post herpetic neuralgia. there are still 2 questions to answer: 1/ do we need to perform the regional anesthesia to relief the pain at an early stage of after no response to the medical treatment? 2/ Are repeated blocks more efficient than a single block?

DETAILED DESCRIPTION:
Study Model:

Randomized prospective registered After approval by the ethical committee of VinMec international Hospitals Institution , after approved registration prior to start the study to www.clinicaltrial.gov, 80 patients will be enrolled to participate to the study.

Inclusion criteria; Acute zona diagnosed by the dermatologist Acute skin rash with blisters in a limited area on one side of the body Eruption Unilateral On dermatome between C5 and S2 Age 18 to 85 years Old [YO], males and females American Society of Anesthesiologists score [ASA] grades I & II Patient who accepted to participate as volunteers and signed an informed consent

Exclusion criteria; Psychiatric disease Central nervous system disease or pre-existing neuropathy Coagulation abnormalities or anti-coagulant treatment (heparins Anti vit K anti thrombin) Contra indication to perform a peripheral nerve block or interfascial block Infection of the skin overlying the puncture site of the block Allergy to local anaesthetic or prednisolone Contra indication to prednisolone ASA III and IV Morbidity Obese BMI > 30 Pregnant woman Baseline evaluation; Date of first rash appeared Pain VAS score from 0 no Pain to 10 the worst imaginable pain Localization of the pain (Skin mapping of the painful area and allodynia area) Quality of life before the rash evaluated by the quality of Life questionnaire SF36 published with a certified translation in Vietnamese As soon as the diagnosis will be done by dermatologist the following treatment will be prescribed according to international published standards of Herpes; Oral administration of Acyclovir 800 mg 5 times a day for 7 days Oral administration of prednisolone except if contra indication 30mg twice daily on d1 > 7 15mg twice daily on d8 > 14 7.5mg twice daily on d15 > 21

Patient flow chart:

Randomization Done by an administrative assistant using a computer program with block randomization.

Group Control = medical treatment with the following pain killers Pain medications Oral administration of Gabapentin 300 mg/d on day 1 and 2 600 mg on day 3 and 4 if pain persists 900 mg on day 5 and 6 if pain persists Oral administration of Paracetamol up to 3 g per day Use of oral narcotic contra-indicated A pain assessment will be done at day 7 if Pain scores < 4 medical treatment will be continued. If Pain score > 4 Patient will be shifted to the group Intervention and will follow the same protocols of this group with randomization done by an administrative assistant using a third computer program table of randomization.

Group Intervention = Early block a second randomization will be done immediately after the first one by an administrative assistant using a second computer program table of randomization.

Single Shot [SS] block : the patient will receive a regional anaesthesia by Inter fascial block, peripheral nerve block. The type of block would be the most appropriate to cover the dermatomes involved in the Herpes according to the mapping done with the higher ration benefit risks. Choice of Block by an anesthesiologist expert in regional anaesthesia techniques. After the block performance if the pain comes back patient will receive the standard medical treatment as in the group medical treatment Repeated [R] Blocks : the patient will receive a regional anaesthesia by Inter fascial block, peripheral nerve block. The type of block would be the most appropriate to cover the dermatomes involved in the Herpes according to the mapping done with the higher ratio benefit risks. The choice of the block will be done by an anesthesiologist expert in regional anaesthesia techniques. The block will be repeated every 48h until the pain will reach VAS < 3 6 h after block recovery.

all the blocks will be performed under US guidance combined if peripheral nerve block or peri plexic block with Neurostimulation guidance to increase the safety of the block performance at the higher level.

The choice of Local anesthetics used will be Ropivacaine 0.5% with the same posology used to performed a regional anaesthesia for surgery.

The patient will be discharged 2 hours after the block performance Follow up

The follow up will be done by :

an pain nurse to analyse VAS at Week 1, 2 and 3 after the inclusion of the patient Satisfaction of patient 0-10 a pain physician to analyse at Month 1, 2 3 and 6 after 1st eruptive sign of Herpes Zona [HZ] eruption development of post herpetic neuralgia defined as Persisting pain beyond the crusting of lesion Pain lasting more than 1, 2 ,3 or 6 months after the acute infection Neuropathic pain with a Douleur Neuropathic 4 [DN4] scale score > 4 DetectPain scale score > 19 Pain level VAS Mapping area of pain to calculate surface Quality of life score at Month 2 3 6 after start of eruptive phase Primary Outcome Quality of pain relief in acute phase VAS score at 1 day / 3 day/ 7 day / 14 Day / 21 day Mapping area surface at day 1, 7 , 14 and 21

Secondary Outcome Development of Neuropathic pain Scale DN4 score > 4 Scale Pain detect Score > 17 Pain intensity Quality of life (QoL) Using the 36 item Short form Health survey [SF36] variation compared to initial assessment

Sample size calculation An estimated 14 patients per group were required to detect a 25% reduction in the mean VAS score in block groups compared to standard treatment group, with a power of 80%, a 2-tailed α of 5%, and a mean VAS-score of 7.25 (SD 1.51) [14] of standard treatment group in the pre-test.

The sample size of 80 patients allowed for a 10% loss to follow-up. Statistical analysis plan Statistical analysis will be performed using STATA 14.0 software. Statistical significant will be set at 5% level (2-tailed). A QoL score will be derived from related variables as stated above, using factor analysis.

Data will be summarized using n (%) for categorical data and median (inter-quartile ranges) for continuous data. Analyses will include Chi-square or Fisher's exact test where appropriate for binomial data. Continuous data will be compared by non-parametric tests.

ELIGIBILITY:
Inclusion Criteria:

* Acute zona diagnosed by the dermatologist

  o Acute skin rash with blisters in a limited area on one side of the body
* Eruption

  * Unilateral
  * On dermatome between C5 and S2
* Age 18 to 85 years old, males and females
* American Society of Anesthesiologists Score [ASA ]grades I & II
* Patient who accepted to participate as volunteers and signed an informed consent

Exclusion Criteria:

* Psychiatric disease
* Central nervous system disease or pre-existing neuropathy
* Coagulation abnormalities or anti-coagulant treatment (heparins Anti vit K anti thrombin)
* Contra indication to perform a peripheral nerve block or interfascial block
* Infection of the skin overlying the puncture site of the block
* Allergy to local anaesthetic or prednisolone
* Contra indication to prednisolone
* ASA III and IV
* Morbidity Obese BMI > 30
* Pregnant woman

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2022-11-12 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity between baseline and the end of treatment | baseline - end of treatment at day 30
  Measure by change in the numeric Visual Analogue Scale (VAS) score. The pain-VAS is a single-item scale which is score from 0 -10. A higher score indicates greater pain intensity (0 = "no pain" and 10 = "worst pain imaginable") 0 is the best score 10 is the worse one

SECONDARY OUTCOMES:
Incidence of postherpetic neuralgia (PHN) after treatment | day 30 - day 60 - day 90 - day 180
  PHN is defined as persisting pain beyond the crusting of cutaneous lesion. Pain lasts more than 1 month after the acute infection with the DN4 scale score > 4 and DetectPain scale score > 19
Chang in quality of life score | Day 1 day 30 - day 60 - day 90 - day 180
  Using the 36-Item Short-Form Health Survey (SF-36) for quality-of-life measurement. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Higher score defines a more favorable health state.
  The overall quality-of-life score at each time-point will be created from all items using an ad-hoc analysis.
The total pain burden during 180 days of follow-up | baseline- every 2 days until day 30 - day 60 - day 90 - day 180
  The total pain burden is quantified using an area-under-the-curve (AUC) method, using the measures of pain intensity and pain duration. Each patient's AUC is calculated as the sum of all areas obtained by multiplying the average of 2 consecutive pain scores by the number of days between the scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Vinmec Health System, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kost RG, Straus SE. Postherpetic neuralgia--pathogenesis, treatment, and prevention. N Engl J Med. 1996 Jul 4;335(1):32-42. doi: 10.1056/NEJM199607043350107. No abstract available. PMID 8637540
- [Background] Galluzzi KE. Management strategies for herpes zoster and postherpetic neuralgia. J Am Osteopath Assoc. 2007 Mar;107(3 Suppl 1):S8-S13. PMID 17488885
- [Background] Pavan-Langston D. Herpes zoster antivirals and pain management. Ophthalmology. 2008 Feb;115(2 Suppl):S13-20. doi: 10.1016/j.ophtha.2007.10.012. PMID 18243927
- [Background] Dworkin RH. Prevention of postherpetic neuralgia. Lancet. 1999 May 15;353(9165):1636-7. doi: 10.1016/S0140-6736(99)00003-3. No abstract available. PMID 10335778
- [Background] Kimberlin DW, Whitley RJ. Varicella-zoster vaccine for the prevention of herpes zoster. N Engl J Med. 2007 Mar 29;356(13):1338-43. doi: 10.1056/NEJMct066061. No abstract available. PMID 17392303
- [Background] Tyring SK. Management of herpes zoster and postherpetic neuralgia. J Am Acad Dermatol. 2007 Dec;57(6 Suppl):S136-42. doi: 10.1016/j.jaad.2007.09.016. PMID 18021865
- [Background] Dworkin RH, Johnson RW, Breuer J, Gnann JW, Levin MJ, Backonja M, Betts RF, Gershon AA, Haanpaa ML, McKendrick MW, Nurmikko TJ, Oaklander AL, Oxman MN, Pavan-Langston D, Petersen KL, Rowbotham MC, Schmader KE, Stacey BR, Tyring SK, van Wijck AJ, Wallace MS, Wassilew SW, Whitley RJ. Recommendations for the management of herpes zoster. Clin Infect Dis. 2007 Jan 1;44 Suppl 1:S1-26. doi: 10.1086/510206. PMID 17143845
- [Background] Schmader KE, Dworkin RH. Natural history and treatment of herpes zoster. J Pain. 2008 Jan;9(1 Suppl 1):S3-9. doi: 10.1016/j.jpain.2007.10.002. PMID 18166460
- [Background] Johnson R. Herpes zoster--predicting and minimizing the impact of post-herpetic neuralgia. J Antimicrob Chemother. 2001 Feb;47 Suppl T1:1-8. doi: 10.1093/jac/47.suppl_1.1. PMID 11160029
- [Background] Schmader KE. Epidemiology and impact on quality of life of postherpetic neuralgia and painful diabetic neuropathy. Clin J Pain. 2002 Nov-Dec;18(6):350-4. doi: 10.1097/00002508-200211000-00002. PMID 12441828
- [Background] Nahm FS, Kim SH, Kim HS, Shin JW, Yoo SH, Yoon MH, Lee DI, Lee YW, Lee JH, Jeon YH, Jo DH. Survey on the treatment of postherpetic neuralgia in Korea; multicenter study of 1,414 patients. Korean J Pain. 2013 Jan;26(1):21-6. doi: 10.3344/kjp.2013.26.1.21. Epub 2013 Jan 4. PMID 23342203
- [Background] Sacks GM. Unmet need in the treatment of postherpetic neuralgia. Am J Manag Care. 2013 Jan;19(1 Suppl):S207-13. PMID 23448093
- [Background] Zhao P, Mei L. A clinical study of paraspinal nerve block on treatment of herpes zoster under ultrasonic guidance. Neurochirurgie. 2019 Dec;65(6):382-386. doi: 10.1016/j.neuchi.2019.06.007. Epub 2019 Jul 23. PMID 31348920
- [Background] Richebe P, Capdevila X, Rivat C. Persistent Postsurgical Pain: Pathophysiology and Preventative Pharmacologic Considerations. Anesthesiology. 2018 Sep;129(3):590-607. doi: 10.1097/ALN.0000000000002238. PMID 29738328
- [Background] Woolf CJ. A new strategy for the treatment of inflammatory pain. Prevention or elimination of central sensitization. Drugs. 1994;47 Suppl 5:1-9; discussion 46-7. doi: 10.2165/00003495-199400475-00003. PMID 7525180
- [Background] Kelly DJ, Ahmad M, Brull SJ. Preemptive analgesia I: physiological pathways and pharmacological modalities. Can J Anaesth. 2001 Nov;48(10):1000-10. doi: 10.1007/BF03016591. PMID 11698320
- [Background] Johnson RW. Consequences and management of pain in herpes zoster. J Infect Dis. 2002 Oct 15;186 Suppl 1:S83-90. doi: 10.1086/342970. PMID 12353192
- [Background] Takeichi H, Watanabe T, Shimojo S. Illusory occluding contours and surface formation by depth propagation. Perception. 1992;21(2):177-84. doi: 10.1068/p210177. PMID 1513667
- [Background] Kumar V, Krone K, Mathieu A. Neuraxial and sympathetic blocks in herpes zoster and postherpetic neuralgia: an appraisal of current evidence. Reg Anesth Pain Med. 2004 Sep-Oct;29(5):454-61. doi: 10.1016/j.rapm.2004.04.010. PMID 15372391
- [Background] Kotani N, Kushikata T, Hashimoto H, Kimura F, Muraoka M, Yodono M, Asai M, Matsuki A. Intrathecal methylprednisolone for intractable postherpetic neuralgia. N Engl J Med. 2000 Nov 23;343(21):1514-9. doi: 10.1056/NEJM200011233432102. PMID 11087880
- [Background] Tekin E, Ahiskalioglu A, Aydin ME, Sengun E, Bayramoglu A, Alici HA. High-thoracic ultrasound-guided erector spinae plane block for acute herpes zoster pain management in emergency department. Am J Emerg Med. 2019 Feb;37(2):375.e1-375.e3. doi: 10.1016/j.ajem.2018.10.028. Epub 2018 Oct 16. PMID 30340986
- [Background] Pasqualucci A, Pasqualucci V, Galla F, De Angelis V, Marzocchi V, Colussi R, Paoletti F, Girardis M, Lugano M, Del Sindaco F. Prevention of post-herpetic neuralgia: acyclovir and prednisolone versus epidural local anesthetic and methylprednisolone. Acta Anaesthesiol Scand. 2000 Sep;44(8):910-8. doi: 10.1034/j.1399-6576.2000.440803.x. PMID 10981565
- [Background] Ji G, Niu J, Shi Y, Hou L, Lu Y, Xiong L. The effectiveness of repetitive paravertebral injections with local anesthetics and steroids for the prevention of postherpetic neuralgia in patients with acute herpes zoster. Anesth Analg. 2009 Nov;109(5):1651-5. doi: 10.1213/ANE.0b013e3181b79075. Epub 2009 Aug 27. PMID 19713253
- [Background] Kim HJ, Ahn HS, Lee JY, Choi SS, Cheong YS, Kwon K, Yoon SH, Leem JG. Effects of applying nerve blocks to prevent postherpetic neuralgia in patients with acute herpes zoster: a systematic review and meta-analysis. Korean J Pain. 2017 Jan;30(1):3-17. doi: 10.3344/kjp.2017.30.1.3. Epub 2016 Dec 30. PMID 28119767
- [Background] Lins L, Carvalho FM. SF-36 total score as a single measure of health-related quality of life: Scoping review. SAGE Open Med. 2016 Oct 4;4:2050312116671725. doi: 10.1177/2050312116671725. eCollection 2016. PMID 27757230
- [Background] BURGOON CF Jr, BURGOON JS, BALDRIDGE GD. The natural history of herpes zoster. J Am Med Assoc. 1957 May 18;164(3):265-9. doi: 10.1001/jama.1957.02980030041010. No abstract available. PMID 13415974
- [Background] HOPE-SIMPSON RE. THE NATURE OF HERPES ZOSTER: A LONG-TERM STUDY AND A NEW HYPOTHESIS. Proc R Soc Med. 1965 Jan;58(1):9-20. doi: 10.1177/003591576505800106. PMID 14267505
- [Background] Eaglstein WH, Katz R, Brown JA. The effects of early corticosteroid therapy on the skin eruption and pain of herpes zoster. JAMA. 1970 Mar 9;211(10):1681-3. No abstract available. PMID 4905733
- [Background] Dworkin RH, Portenoy RK. Proposed classification of herpes zoster pain. Lancet. 1994 Jun 25;343(8913):1648. doi: 10.1016/s0140-6736(94)93106-2. No abstract available. PMID 7911959
- [Background] Riopelle JM, Naraghi M, Grush KP. Chronic neuralgia incidence following local anesthetic therapy for herpes zoster. Arch Dermatol. 1984 Jun;120(6):747-50. PMID 6721540
- [Result] Bennett GJ, Watson CP. Herpes zoster and postherpetic neuralgia: past, present and future. Pain Res Manag. 2009 Jul-Aug;14(4):275-82. doi: 10.1155/2009/380384. PMID 19714266